CLINICAL TRIAL: NCT01874093
Title: A Multi-center, Rand., Double Blind, Sham Control, Parallel Arm Post Mech. Thrombectomy and/or rtPA Trial to Assess Safety and Effectiveness of the Ischemic Stroke System, as an Adjunct to Stand. of Care in Subjects With Acute Isch. Stroke
Brief Title: IMPACT- 24Bt Post Mech. Thrombectomy and/or rtPA TRIAL IMPlant Augmenting Cerebral Blood Flow 24 Hours From Stroke Onset
Acronym: IMPACT-24Bt
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLP1050035
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2017-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Stimulation (Experimental): INS implantation, 5 Days of Ischemic Stroke System (ISS) Stimulation + Standard of Care
  Interventions: Device: The Ischemic Stroke System
- Sham Stimulation (Sham Comparator): Sham implantation, 5 Days of Sham Stimulation + Standard of Care
  Interventions: Device: Sham control

INTERVENTIONS:
Device: The Ischemic Stroke System — SPG stimulation and standard of care
  Arms: Active Stimulation
Device: Sham control — Sham stimulation and standard of care
  Arms: Sham Stimulation

SUMMARY:
The primary objective of the study is to assess the safety and effectiveness of SPG stimulation with the ISS in a 24 hour window, in patients with an acute ischemic stroke in the anterior circulation, who received Mechanical Thrombectomy and/or IV-rtPA and Standard of Care.

DETAILED DESCRIPTION:
This will be a multi-center, multinational, randomized, double blind, sham control, adjunctive to Standard of Care, parallel arm study and will include ongoing DSMB review of accumulated safety data.

The study has three phases:

Phase I - Implantation Safety Assessment

* Number of patients: 20 (at least 10 implantations)
* Implanters: only certified implanters who already performed implantation of ISS in previous studies
* Continue to the next phase if there are no serious procedure complications related to IV-rtPA (as determined by the implanter). Otherwise, implement retirements and continue only after DSMB approval.

DSMB meetings: after 10 implantations

Phase II - Symptomatic Intracranial Hemorrhage Assessment (sICH):

* Number of patients: 50 (additional 30)
* Implanters: all certified implanters
* Verify no clinically meaningful difference between treated and control. A clinically meaningful difference is a difference of more than 3 sICH cases within the first 5 days of treatment, in the treated arm compared to the control arm.

In case of clinically meaningful difference, implement retirements.

* Continue to phase III after DSMB approval.
* DSMB meetings: after 30 and 50 patients

Phase III - Entire study population, DSMB meetings at 100 and 150 patients

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 40 years and ≤ 80 years for male and 85 for female subjects
2. Clinical diagnosis of an acute ischemic stroke in the Carotid, Middle or Anterior Cerebral Artery territories based on general physical examination and neurological examination.
3. Imaging findings demonstrating signs of ischemia (or total arterial occlusion prior to the MT procedure) in the anterior circulation, consistent with the clinical diagnosis.
4. Performance of MT within <8 hours from stroke onset and/or administration of IV-rtPA within ≤ 4.5 hours from stroke onset.
5. NIHSS ≥ 7 and ≤ 18 within 2 hours prior to implantation.
6. Ability to initiate treatment within

   ≤ 24 hours from stroke onset.
7. Signed informed consent from patient him/herself or legally authorized representative if applicable.

Exclusion Criteria:

1. Neuro-imaging evidence of any intracranial hemorrhage (including suspect of Sub Arachnoid Hemorrhage) or hemorrhagic transformation of brain infarct or other significant abnormality (e.g. tumor, abscess)
2. Massive stroke, defined as acute parenchymal lesion with effacement of cerebral sulci in over 2/3 of the MCA territory.
3. Acute stroke due to lacunar infarct as defined by a clinical syndrome (pure motor hemiparesis, ataxic hemiparesis, sensorimotor stroke, dysarthria-clumsy hand syndrome), unless brain imaging demonstrates a relevant lesion > 1.5 cm in size.
4. Clinical signs and symptoms or evidence for a relevant lesion by neuro-imaging of an acute ischemic stroke in the posterior circulation (Vertebral, Basilar and/or Posterior Cerebral Artery territories), including but not limited to brain-stem findings and/or cerebellar findings and/or isolated homonymous hemianopia or cortical blindness.
5. Minor stroke with non-disabling deficit or rapidly improving neurological symptoms.
6. Clinical signs and symptoms or imaging evidence of bilateral stroke.
7. Treated with IA-rtPA for the current stroke.
8. Complicated MT procedure (including procedures with more than 3 clot removal attempts (catheter passes), or MT procedure that lasted more than 2 hours)
9. NIHSS level of consciousness score ≥ 2.
10. Previous stroke in the last 6 months or previous stroke with existing sequelae or with mRS > 0 for any reason
11. Pre-existing disability; Pre-existing Modified Rankin Score >1, even if not stroke-related.
12. Patients with bleeding propensity and/or one of the following: INR≥ 1.8, prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec., platelets count < 75×109/L prior to the implantation/sham procedure.
13. Known cerebral arteriovenous malformation, cerebral aneurysm.
14. Seizure at onset.
15. Blood glucose concentration < 60 mg/dL.
16. Clinical suspicion of septic embolus.
17. Uncontrolled hypertension (systolic >185 mmHg and/or diastolic >110 mmHg), demonstrated on each of three repeated measurements taken within one hour regardless of whether or not the patient is taking antihypertensive medications.
18. Serious systemic infection.
19. Women known to be pregnant or having a positive or indeterminate pregnancy test.
20. Patients with other implanted neural stimulator/ electronic devices (pacemakers, etc.).
21. History of SPG ablation ipsilateral to the stroke side.
22. Any condition in the oral cavity that prevents implantation of the INS, such as patient is intubated, orthodontics or non-hygienic condition.
23. Life expectancy < 1 year from causes other than stroke.
24. Participating in any other therapeutic investigational trial within the last 30 days.
25. Known sensitivity to any medication to be used during study.
26. Subjects who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Conditions may include: cardiovascular, vascular, pulmonary, hepatic, renal or neurological (other than acute ischemic stroke), or neoplastic diseases, as determined by medical history, physical examination, laboratory tests, or ECG.
27. Subjects who, in the judgment of the investigator, are likely to be non-compliant or uncooperative during the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-05; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Distribution of patients across the ordinal modified Rankin scale (mRS) | 90 days
  The primary effectiveness endpoint will be the modified Rankin Scale (mRS) evaluated by the site on Day 90±7.
  The statistical analysis of the primary effectiveness endpoint will be: Sliding Dichotomous mRS.

SECONDARY OUTCOMES:
Distribution of patients with NIHSS best language score ≥ 2 at screening across the ordinal modified Rankin scale (mRS) | 90 days
  The secondary effectiveness endpoint will be the modified Rankin Scale (mRS) evaluated by the site on Day 90±7 for patients with NIHSS best language score ≥ 2 at screening.
  The statistical analysis of the primary effectiveness endpoint will be: Sliding Dichotomous mRS.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shai, Study Director — BrainsGate
Locations (1):
- Vall d'Hebron, Barcelona, Spain